CLINICAL TRIAL: NCT02084498
Title: A Randomized Controlled Large Study of Flexible Intensified Insulin Therapy (FIIT) With Carbohydrate Counting (CHC) Versus FIIT With Carbohydrate Counting and Automated Bolus Calculation (ABC)
Brief Title: Advanced Carbohydrate Counting and Automated Bolus Calculation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Eva Hommel, Senior Consultant, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StenoABC
Record Dates: First submitted 2014-02-24; First posted 2014-03-12 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Type 1 Diabetes
Keywords: Automated bolus calculator (ABC); Advanced carbohydrate counting (ACC); Patient empowerment
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACC (Active Comparator): Training in advanced carbohydrate counting
  Interventions: Behavioral: Advanced Carbohydrate Counting
- ACC + ABC (Experimental): Training in advanced carbohydrate counting plus the use of an automated bolus calculator.
  Interventions: Device: Automated bolus calculator; Behavioral: Advanced Carbohydrate Counting

INTERVENTIONS:
Device: Automated bolus calculator — Training in Advanced Carbohydrate Counting and the use of an automated bolus calculator according to the BolusCal concept.
  Other Names: Accu-Chek Aviva Expert, Roche Diagnostics
  Arms: ACC + ABC
Behavioral: Advanced Carbohydrate Counting — Training in advanced carbohydrate counting.

SUMMARY:
The investigators hypothesize, that non-optimally treated carbohydrate counting-naïve patients with type 1 diabetes can achieve better metabolic control by counting carbohydrates, and that the metabolic control can be further improved with concurrent use of Accu-Chek Aviva Expert. Additionally, the investigators propose that carbohydrate counting will lead to better quality of life as a result of fewer restrictions when eating and less variation in blood glucose. Finally the investigators hypothesize that the use of Accu-Chek Aviva Expert will lead to fewer hypoglycemic episodes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes
* Age >18 years
* Diabetes duration more than 12 months
* Multiple Daily Injections therapy (fast acting analog for meals; long acting analog as basal)
* HbA1c between 8.0% and 11.3%

Exclusion Criteria:

* Present or former practice of carbohydrate counting
* Gastroparesis
* Pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2012-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Baseline, 12 months

SECONDARY OUTCOMES:
Frequency of serious hypoglycemic events | Baseline, 12 months

OTHER OUTCOMES:
Frequency of glucose below, in or above target 4-8 mmol/l assessed by blinded Continuous Glucose Monitoring 6 days before study start and 6 days before ending the study | Baseline, 12 months
Frequency of blood glucose measurements assessed by meter download before randomization and at each visit during the study | Baseline, 12 months
Treatment Satisfaction | Baseline, 12 months
  Measured by Diabetes Treatment Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eva E Hommel, MD, DMSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Background] Schmidt S, Meldgaard M, Serifovski N, Storm C, Christensen TM, Gade-Rasmussen B, Norgaard K. Use of an automated bolus calculator in MDI-treated type 1 diabetes: the BolusCal Study, a randomized controlled pilot study. Diabetes Care. 2012 May;35(5):984-90. doi: 10.2337/dc11-2044. Epub 2012 Feb 16. PMID 22344610
- [Derived] Hommel E, Schmidt S, Vistisen D, Neergaard K, Gribhild M, Almdal T, Norgaard K. Effects of advanced carbohydrate counting guided by an automated bolus calculator in Type 1 diabetes mellitus (StenoABC): a 12-month, randomized clinical trial. Diabet Med. 2017 May;34(5):708-715. doi: 10.1111/dme.13275. Epub 2016 Nov 10. PMID 27761942